CLINICAL TRIAL: NCT05671588
Title: Cardiovascular Fitness and the Influence of a Controlled Combined Exercise Program on Fatigue and Depression of Newly Diagnosed Patients With Multiple Sclerosis
Brief Title: Cardiovascular Fitness of Patients With Multiple Sclerosis, Effect of Exercise on Fatigue and Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01/RVO-FNOs/2022; 01/RVO-FNOs/2022 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2022-12-12; First posted 2023-01-04 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Controlled combined exercise; Cardiovascular fitness; Fatigue; Depression
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Depression

STUDY DESIGN:
Intervention Model Description: The study subjects will be enrolled into two parallel groups.
Who Masked: Outcomes Assessor
Masking Description: All participants of the study will undergo a clinical examination including a questionnaire survey and spiroergometry - examiners will not have access to intervention documents before and after the intervention (period of 6 months), as well as examiners will not perform the therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Controlled combined program (aerobic-resistant) (Experimental): Patients randomized into the Experimental arm will undergo controlled exercise on a cycling ergometer in combination with strength training on a multifunctional fitness device for 1-hour duration, twice a week for one month, and once a week for the next month (12 therapies in total).
  Interventions: Procedure: Controlled combined exercise group
- Conventional rehabilitation (Active Comparator): Patients randomized into this study arm will undergo conventional rehabilitation.
  Interventions: Procedure: Conventional rehabilitation
- No intervention (No Intervention): Patients randomized into this study arm will undergo no intervention and will serve as the control group.

INTERVENTIONS:
Procedure: Controlled combined exercise group — Patients will undergo protocol-defined combined aerobic-resistant therapy on a cycling ergometer and multifunctional fitness device
  Arms: Controlled combined program (aerobic-resistant)
Procedure: Conventional rehabilitation — Patients will undergo conventional rehabilitation.
  Arms: Conventional rehabilitation

SUMMARY:
This study is focused on patients with multiple sclerosis (MS), their cardiovascular fitness, and the effect of combined controlled training on the perception of fatigue, the development of depression, and quality of life in the first year after diagnosis.

DETAILED DESCRIPTION:
The main goal is to find out if fatigue, depression, and quality of life depend on the type of training as well as controlled management of newly diagnosed patients. Fatigue is one of the frequent disabling symptoms and the most difficult to influence pharmacologically. It could lead to inactivity and the progression of deconditioning. We know from systematic reviews that aerobic activity leads to improvement in fatigue, however, there are also opinions about exercise intolerance due to disruption of cardiac autonomy control. The investigators will try to determine whether early rehabilitation intervention leads to support and motivation of patients with an incurable chronic neurodegenerative disease to improve the patient condition and contentment. The researchers will focus on effective training by comparing the study group with a control group of patients undergoing conventional rehabilitation versus a protocol-defined controlled combined (aerobic-resistant) exercise program - based on the results of spiroergometry. Both groups will be treated at ambulatory sections by protocol-defined rehabilitation for a 1-hour duration, twice a week for one month, and once a week for the next month (12 therapies in total). The control group will be educated in exercises according to kinesiological analysis to do regularly at home. Finally, the researchers will see if early intervention leads to a change in the active approach of probands.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 45 years
* Newly diagnosed patients with multiple sclerosis
* Relapsing-remitting MS (RRMS) or clinically isolated syndrome (CIS)
* EDSS 0-6
* Signed informed consent

Exclusion Criteria:

* Progressive forms of MS (PRMS or SPMS), Malignant MS
* Non-cooperation, disagreement with the study
* Contraindication to spiroergometry

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal aerobic capacity (VO2max.kg-1) | 6 months
  Change after six months follow up in conventional, experimental and control group
Power to weight ratio (W.kg-1) | 6 months
  Change after six months follow up in conventional, experimental and control group

SECONDARY OUTCOMES:
Modified Fatigue Impact Scale (MFIS) | 6 months
  Self-reported measure of level of fatigue, minimum 0 points, maximum 84 points - the less score means less fatigue
Symptom-Checklist-90-Standard (SCL-90-S) | 6 months
  Change in result of percentile score
Beck Depression Inventory Score II (BDI II) | 6 months
  Self-reported rating inventory that measures characteristic attitudes and symptoms of depression, 0-13 - minimal or none depression, 29-63 - severe depression
36-Item Short Form Survey (SF-36) | 6 months
  Self-reported measure of health-related quality of life, minimum 0 points, maximum 100 points - the higher score is the sign of better quality of life
Maximal heart rate (bpm) | 6 months
  Change after six months follow up in conventional, experimental and control group
Heart rate variability (ms) | 6 months
  Change after six months follow up in conventional, experimental and control group
Body composition analysis %) | 6 months
  Body composition (fat, water, muscle, bone mass) analysis will be performed in study subjects and expressed as per cent.

OTHER OUTCOMES:
Cost-benefit analysis of early rehabilitation intervention (CZK) | 6 months
  Cost-benefit analysis of early rehabilitation intervention will be performed and expressed as the price in Czech crowns (CZK).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Šilarová, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] Razazian N, Kazeminia M, Moayedi H, Daneshkhah A, Shohaimi S, Mohammadi M, Jalali R, Salari N. The impact of physical exercise on the fatigue symptoms in patients with multiple sclerosis: a systematic review and meta-analysis. BMC Neurol. 2020 Mar 13;20(1):93. doi: 10.1186/s12883-020-01654-y. PMID 32169035
- [Background] Taul-Madsen L, Connolly L, Dennett R, Freeman J, Dalgas U, Hvid LG. Is Aerobic or Resistance Training the Most Effective Exercise Modality for Improving Lower Extremity Physical Function and Perceived Fatigue in People With Multiple Sclerosis? A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2021 Oct;102(10):2032-2048. doi: 10.1016/j.apmr.2021.03.026. Epub 2021 Apr 24. PMID 33901439
- [Background] Cruickshank TM, Reyes AR, Ziman MR. A systematic review and meta-analysis of strength training in individuals with multiple sclerosis or Parkinson disease. Medicine (Baltimore). 2015 Jan;94(4):e411. doi: 10.1097/MD.0000000000000411. PMID 25634170
- [Background] Hansen D, Wens I, Keytsman C, Eijnde BO, Dendale P. Is long-term exercise intervention effective to improve cardiac autonomic control during exercise in subjects with multiple sclerosis? A randomized controlled trial. Eur J Phys Rehabil Med. 2015 Apr;51(2):223-31. Epub 2014 Mar 6. PMID 24603938